CLINICAL TRIAL: NCT04726969
Title: Efficacy and Safety of Combination Moxidectin and Albendazole, Ivermectin and Albendazole and Albendazole Alone in Adolescents and Adults Infected With Trichuris Trichiura: a Randomized Controlled Trial
Brief Title: Efficacy and Safety of MOX/ALB Co-administration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jennifer Keiser (Other)
Collaborators: Centre Suisse de Recherches Scientifiques en Cote d'Ivoire (Other)
Responsible Party: Sponsor-Investigator, Jennifer Keiser, Prof. Dr., Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MAC_CI_1
Record Dates: First submitted 2021-01-18; First posted 2021-01-27 (Actual); Results first posted 2023-02-02 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Trichuriasis; Ascariasis; Hookworm Infections
Keywords: Albendazole; Moxidectin; Ivermectin; Anthelmintics; T. trichiura; A. lumbricoides; Hookworm; Whipworm; Soil-transmitted helminths
MeSH Terms: conditions — Trichuriasis; Ascariasis; Hookworm Infections; Ancylostomiasis | interventions — moxidectin; Tablets; Albendazole; Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The parallel group trial co-administered moxidectin/albendazole versus albendazole alone will be double blinded (i.e. study participants and the trial team/researchers conducting the treatment and assessing the outcomes will be blinded) using tablets including appearance-matched placebos, while the ivermectin/albendazole arm will be open label due to the nature of ivermectin (i.e. requiring bodyweight-dependent doses).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm A: moxidectin and albendazole (Experimental): Combination therapy of moxidectin (8 mg, i.e. 4 tablets of 2 mg) and albendazole (Zentel®, 1 tablet of 400 mg) administered orally at day 0
  Interventions: Drug: Moxidectin 2 mg Oral Tablet; Drug: Albendazole 400 mg Oral Tablet
- Arm B: albendazole (Placebo Comparator): Placebo (for moxidectin, 4 tablets) and albendazole (Zentel®, 1 tablet of 400 mg) administered orally at day 0
  Interventions: Drug: Albendazole 400 mg Oral Tablet
- Arm C: ivermectin and albendazole (Experimental): Combination therapy of ivermectin (Stromectol®, 200 µg/kg using tablets of 3 mg) and albendazole (Zentel®, 1 tablet of 400 mg) administered orally at day 0
  Interventions: Drug: Albendazole 400 mg Oral Tablet; Drug: Ivermectin 3 mg Oral Tablet

INTERVENTIONS:
Drug: Moxidectin 2 mg Oral Tablet — Tablets of 2 mg moxidectin
  Arms: Arm A: moxidectin and albendazole
Drug: Albendazole 400 mg Oral Tablet — Tablets of 400 mg albendazole
  Other Names: Zentel®
Drug: Ivermectin 3 mg Oral Tablet — Tablets of 3 mg ivermectin
  Other Names: Stromectol®
  Arms: Arm C: ivermectin and albendazole

SUMMARY:
This study is a double-blind randomized controlled superiority trial aiming at providing evidence on the efficacy and safety of co-administered moxidectin and albendazole versus albendazole monotherapy (standard of care) against whipworm (T. trichiura) infections in adolescents and adults (12-60 years) in Côte d'Ivoire. One arm of patients will be treated with albendazole-ivermectin.

As measure of efficacy of the treatment the cure rate (percentage of egg-positive subjects at baseline who become egg-negative after treatment) will be determined 14-21 days post-treatment.

DETAILED DESCRIPTION:
This study is a double-blind randomized clinical trial which aims at providing evidence on the efficacy and safety of co-administered moxidectin and albendazole versus albendazole monotherapy (standard of care) against T. trichiura infections in adolescents and adults (12-60 years) in Côte d'Ivoire. Additionally, this study aims to substantiate evidence on the efficacy and safety of co-administered ivermectin and albendazole compared to albendazole monotherapy against T. trichiura in the same age group.

The primary objective of the trial is to comparatively assess the efficacy in terms of cure rate (CR) against T. trichiura infections among adolescents and adults (aged 12 to 60 years) of moxidectin/albendazole combination therapy and albendazole monotherapy.

The secondary objectives of the trial are to compare the egg reduction rates (ERR) of these treatment regimens (moxidectin/albendazole combination therapy vs. albendazole monotherapy) against T. trichiura, to assess the CRs and ERRs in T. trichiura-infected participants given ivermectin/albendazole combination therapy compared to those given albendazole monotherapy, to determine the CRs and ERRs of the drugs in study participants co-infected with A. lumbricoides and hookworm, and to evaluate the safety and tolerability of the treatment regimens. In addition, this study aims to characterize population pharmacokinetics and drug-drug interactions of the study drugs albendazole and ivermectin in T. trichiura infected adolescents (aged 12 to 20 years), to evaluate pharmacogenomics of ivermectin using whole genome sequencing, and to assess the effect of the gut microbiota on pharmacokinetics parameters and treatment outcome (CRs and ERRs), and drug-specific off-target effects of anthelmintic treatment on gut microbial communities in post-treatment samples.

After obtaining informed consent from individual/parents and/or caregivers, the medical history of the participants will be assessed with a standardized questionnaire, in addition to a clinical examination carried out by the study physician before treatment. Enrollment will be based on two stool samples, which will be collected, if possible, on two consecutive days or otherwise within a maximum of 5 days. All stool samples will be examined with duplicated Kato-Katz thick smears by experienced laboratory technicians.

Randomization of participants into the three treatment arms will be stratified according to intensity of infection. All participants will be interviewed before treatment, 3 and 24 hours and 14-21 days after treatment about the occurrence of adverse events. The efficacy of the treatment will be determined 14-21 days post-treatment by collecting another two stool samples.

The primary analysis will include all participants with primary end point data (available case analysis). Supplementary, a per-protocol analysis will be conducted. CRs will be calculated as the percentage of egg-positive subjects at baseline who become egg-negative after treatment. Differences among CRs between treatment arms will be analysed using crude and adjusted logistic regression modeling (adjustment for age, sex and weight).

Geometric and arithmetic mean egg counts will be calculated for the different treatment arms before and after treatment to assess the corresponding ERRs.

Bootstrap resampling method with 5,000 replicates will be used to calculate 95% confidence intervals (CIs) for differences in ERRs.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 12 and 60 years
* Written informed consent signed by either parents/caregivers for underage adolescents (aged 12-17 years) or by the participant him/herself (18-60 years of age); and written assent by underage participant
* Agree to comply with study procedures, including provision of two stool samples at the beginning (baseline) and at follow-up assessment 14-21 days after treatment
* Willing to be examined by a study physician prior to treatment
* At least two slides of the quadruple Kato-Katz thick smears positive for T. trichiura and infection intensities of at least 48 EPG

Exclusion Criteria:

* Presence or signs of major systemic illnesses, e.g. body temperature ≥ 38°C, severe anemia (below 80g/l Hb according to WHO) upon initial clinical assessment
* Known or suspected infection with Loa loa
* History of acute or severe chronic disease
* Abnormal liver function assessed by multiple biochemical blood-based analyses
* Recent use of anthelmintic drug (within past 4 weeks)
* Attending other clinical trials during the study
* Pregnancy, lactating, and/or planning to become pregnant within the next 3 months
* Known allergy to study medications (i.e. albendazole, ivermectin or moxidectin)
* Taking medication with known contraindication to or interaction with study drugs

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 255 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Suisse de Recherches Scientifiques en Côte d'Ivoire (CSRS), Abidjan, Côte d’Ivoire

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sprecher VP, Coulibaly JT, Hurlimann E, Hattendorf J, Keiser J. Efficacy and Safety of Moxidectin-Albendazole and Ivermectin-Albendazole Combination Therapy Compared to Albendazole Monotherapy in Adolescents and Adults Infected with Trichuris trichiura: A Randomized, Controlled Superiority Trial. Clin Infect Dis. 2023 Nov 11;77(9):1294-1302. doi: 10.1093/cid/ciad387. PMID 37357904

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: Moxidectin and Albendazole | Arm B: Albendazole | Arm C: Ivermectin and Albendazole
Started | 85 | 84 | 86
Completed | 72 | 67 | 71
Not Completed | 13 | 17 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Moxidectin and Albendazole | Arm B: Albendazole | Arm C: Ivermectin and Albendazole | Total
Number analyzed (Participants) | 85 | 84 | 86 | 255
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 38 | 39 | 33 | 110
  Between 18 and 65 years | 47 | 45 | 53 | 145
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.1 (16.1) | 26.7 (14.5) | 29.9 (15.4) | 28.9 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 49 | 137
  Male | 41 | 40 | 37 | 118
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Côte D'Ivoire | 85 | 84 | 86 | 255

OUTCOME MEASURES:

1. Primary Outcome: Cure Rate (CR) of Moxidectin/Albendazole Combination Therapy Compared to Albendazole Monotherapy Against T. Trichiura
Description: The CR will be calculated as the proportion of participants converting from being egg positive pre-treatment to egg negative post-treatment, multiplied by 100.
Time Frame: 14-21 days after treatment
Population: Available case analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants (%)
Arm/Group | Arm A: Moxidectin and Albendazole | Arm B: Albendazole
Number analyzed (Participants) | 72 | 67
percentage of participants (%) | 15.3 [7.9 to 25.7] | 13.4 [6.3 to 24.0]

2. Secondary Outcome: Egg Reduction Rate (ERR) of Moxidectin/Albendazole Combination Therapy Compared to Albendazole Monotherapy Against T. Trichiura
Description: Eggs per gram of stool (EPG) will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. Geometric and arithmetic mean egg counts will be calculated for the two treatment arms before and after treatment to assess the corresponding ERRs.
Time Frame: 14-21 days after treatment
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Arm A: Moxidectin and Albendazole | Arm B: Albendazole
Number analyzed (Participants) | 72 | 67
percent change | 67.0 [47.8 to 80.1] | 60.2 [35.7 to 76.5]

3. Secondary Outcome: Cure Rate (CR) of Ivermectin/Albendazole Combination Therapy Compared to Albendazole Monotherapy Against T. Trichiura
Description: as for outcome 1
Time Frame: 14-21 days after treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants (%)
Arm/Group | Arm B: Albendazole | Arm C: Ivermectin and Albendazole
Number analyzed (Participants) | 67 | 71
percentage of participants (%) | 13.4 [6.3 to 24.0] | 22.5 [13.5 to 34.0]

4. Secondary Outcome: Egg Reduction Rate (ERR) of Ivermectin/Albendazole Combination Therapy Compared to Albendazole Monotherapy Against T. Trichiura
Description: as for outcome 2
Time Frame: 14-21 days after treatment
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Arm B: Albendazole | Arm C: Ivermectin and Albendazole
Number analyzed (Participants) | 67 | 71
percent change | 60.2 [35.7 to 76.5] | 81.5 [68.8 to 89.1]

5. Secondary Outcome: Cure Rates (CRs) of the Study Drugs Against Ascaris Lumbricoides Infections in Co-infected Participants
Description: as for outcome 1
Time Frame: 14-21 days after treatment
Population: Available case analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants (%)
Arm/Group | Arm A: Moxidectin and Albendazole | Arm B: Albendazole | Arm C: Ivermectin and Albendazole
Number analyzed (Participants) | 22 | 22 | 33
percentage of participants (%) | 95.5 [86.0 to 100] | 95.5 [86.0 to 100] | 100 [100 to 100]

6. Secondary Outcome: Egg Reduction Rates (ERRs) of the Study Drugs Against Ascaris Lumbricoides Infections in Co-infected Participants
Description: Eggs per gram of stool (EPG) will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. Geometric and arithmetic mean egg counts will be calculated for the three treatment arms before and after treatment to assess the corresponding ERRs.
Time Frame: 14-21 days after treatment
Population: Available case analysis
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Arm A: Moxidectin and Albendazole | Arm B: Albendazole | Arm C: Ivermectin and Albendazole
Number analyzed (Participants) | 22 | 22 | 33
percent change | 100 [100 to 100] | 100 [100 to 100] | 100 [100 to 100]

7. Secondary Outcome: Cure Rates (CRs) of the Study Drugs Against Hookworm Infections in Co-infected Participants
Description: as for outcome 1
Time Frame: 14-21 days after treatment
Population: Available case analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants (%)
Arm/Group | Arm A: Moxidectin and Albendazole | Arm B: Albendazole | Arm C: Ivermectin and Albendazole
Number analyzed (Participants) | 1 | 8 | 5
percentage of participants (%) | 100 [100 to 100] | 37.5 [0 to 80.8] | 20.0 [0 to 75.5]

8. Secondary Outcome: Egg Reduction Rates (ERRs) of the Study Drugs Against Hookworm Infections in Co-infected Participants
Description: as for outcome 6
Time Frame: 14-21 days after treatment
Population: Available case analysis
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Arm A: Moxidectin and Albendazole | Arm B: Albendazole | Arm C: Ivermectin and Albendazole
Number analyzed (Participants) | 1 | 8 | 5
percent change | 100 [100 to 100] | 95.7 [78.5 to 99.3] | 90.7 [78.6 to 97.7]

9. Secondary Outcome: Number of Participants Reporting Adverse Events (AEs)
Description: Participants will be monitored at the site for 3 hours following treatment for any acute AEs and reassessment will be done at 24h post-treatment. In addition, participants will be interviewed 3 and 24 hours after treatment and retrospectively at days 14-21 about the occurrence of AEs.
Time Frame: 3 hours, 24 hours and 14-21 days after treatment
Population: Analysis population at 3 hours after drug administration: N=255 Analysis population at 24 hours after drug administration: N=250 Analysis population at 14-21 days after drug administration: N=210
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Moxidectin and Albendazole | Arm B: Albendazole | Arm C: Ivermectin and Albendazole
Number analyzed (Participants) | 85 | 84 | 86
Participants
  3 hours: Headache | 1 | 5 | 7
  3 hours: Abdominal pain | 4 | 6 | 8
  3 hours: Nausea | 3 | 2 | 2
  3 hours: Diarrhea | 2 | 1 | 1
  3 hours: Itching | 1 | 6 | 2
  3 hours: Symptoms related to immune system activation | 3 | 5 | 5
  24 hours: Headache: number analyzed (Participants) | 84 | 82 | 84
  24 hours: Headache | 4 | 9 | 6
  24 hours: Abdominal pain: number analyzed (Participants) | 84 | 82 | 84
  24 hours: Abdominal pain | 8 | 5 | 12
  24 hours: Nausea: number analyzed (Participants) | 84 | 82 | 84
  24 hours: Nausea | 1 | 0 | 3
  24 hours: Diarrhea: number analyzed (Participants) | 84 | 82 | 84
  24 hours: Diarrhea | 5 | 4 | 7
  24 hours: Itching: number analyzed (Participants) | 84 | 82 | 84
  24 hours: Itching | 9 | 8 | 4
  24 hours: Symptoms related to immune system activation | 1 | 5 | 3
  14-21 days: Headache: number analyzed (Participants) | 72 | 67 | 71
  14-21 days: Headache | 0 | 0 | 0
  14-21 days: Abdominal pain: number analyzed (Participants) | 72 | 67 | 71
  14-21 days: Abdominal pain | 0 | 0 | 0
  14-21 days: Nausea: number analyzed (Participants) | 72 | 67 | 71
  14-21 days: Nausea | 0 | 0 | 0
  14-21 days: Diarrhea: number analyzed (Participants) | 72 | 67 | 71
  14-21 days: Diarrhea | 0 | 0 | 0
  14-21 days: Itching: number analyzed (Participants) | 72 | 67 | 71
  14-21 days: Itching | 0 | 0 | 0
  14-21 days: Symptoms related to immune system activation | 0 | 0 | 0

10. Other Pre Specified Outcome: Concentrations of Albendazole and Ivermectin/Albendazole Combination in Adolescents (Aged 12 to 20 Years)
Description: For characterization of population pharmacokinetics (PK) and drug-drug interaction parameters ivermectin, albendazole and its metabolites will be quantified using a validated liquid chromatography tandem mass spectrometry (LC-MS/MS) method. Drug concentrations will be calculated by interpolation from a calibration curve with a lower limit of quantification of 1-5 ng/ml.
Time Frame: 0 to 24 hours after treatment
Population: Arm B did not receive ivermectin, thus no concentration was measured.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Arm B: Albendazole | Arm C: Ivermectin and Albendazole
Number analyzed (Participants) | 8 | 8
ng/ml
  cmax (albendazole) [ng/ml] | 26.5 [20.0 to 36.8] | 26.5 [20.0 to 36.8]
  cmax (ivermectin) [ng/ml]: number analyzed (Participants) | 0 | 8
  cmax (ivermectin) [ng/ml] |  | 40.1 [32.4 to 59.1]

11. Other Pre Specified Outcome: Genetic Variants in Ivermectin/Albendazole Participants
Description: In case of unexpected results for outcome measure 10 (Concentrations of Albendazole and Ivermectin/Albendazole Combination in Adolescents (Aged 12 to 20 Years)), whole genome sequencing will be performed on blood samples from participants in the ivermectin/albendazole arm to analyse genetic variation of relevance for ivermectin metabolism.
Time Frame: before treatment, i.e. at enrolment
Population: This analysis has not been performed.
Arm/Group | Arm C: Ivermectin and Albendazole
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Gut Bacterial Communities in Stool Samples
Description: Taxonomic relative abundances of gut bacterial communities will be analysed with high-throughput sequencing. Absolute abundances of specific taxa will be measured using taxon-specific qPCR. Changes in relative and absolute abundances will be measured before and after treatment.
Time Frame: before treatment, i.e. at screening, and 14-21 days after treatment
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Exploratory Outcome: Number of Participants Within Each Blood Type Category (A, B, AB and 0)
Description: Blood type of participants will be collected during clinical examination prior treatment using blood type determination cards.
Time Frame: before treatment, i.e. at enrolment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Moxidectin and Albendazole | Arm B: Albendazole | Arm C: Ivermectin and Albendazole
Number analyzed (Participants) | 85 | 84 | 86
Participants
  Blood type 0 | 48 | 47 | 47
  Blood type A | 20 | 18 | 12
  Blood type B | 15 | 16 | 24
  Blood type AB | 2 | 3 | 3

ADVERSE EVENTS:
Time Frame: 14-21 days
Description: Participants were monitored at the site for 3 hours following treatment for any acute adverse events and reassessment was done at 24 hours post-treatment. In addition, participants will be interviewed 3 and 24 hours after treatment and retrospectively at days 14-21 about the occurrence of AEs.
Arm/Group | Arm A: Moxidectin and Albendazole | Arm B: Albendazole | Arm C: Ivermectin and Albendazole
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/84 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/84 | 0/86
Other Adverse Events (participants affected / at risk) | 31/85 | 26/84 | 34/86
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Moxidectin and Albendazole (N=85) | Arm B: Albendazole (N=84) | Arm C: Ivermectin and Albendazole (N=86)
Headache (General disorders) | 4 (5) | 12 (14) | 12 (13)
Abdominal pain (Gastrointestinal disorders) | 11 (12) | 10 (11) | 18 (20)
Nausea (General disorders) | 4 (4) | 2 (2) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 6 (7) | 4 (5) | 7 (8)
Itching (Skin and subcutaneous tissue disorders) | 9 (10) | 11 (14) | 5 (6)
Allergic reaction (General disorders) | 2 (2) | 0 (0) | 2 (2)
Symptoms related to immune system activation (Immune system disorders) | 4 (4) | 10 (10) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/69/NCT04726969/Prot_SAP_000.pdf